CLINICAL TRIAL: NCT02255656
Title: A Long-term Follow-up Study for Multiple Sclerosis Patients Who Have Completed the Alemtuzumab Extension Study (CAMMS03409)
Brief Title: Phase IIIB-IV Long-Term Follow-up Study for Patients Who Participated in CAMMS03409
Acronym: TOPAZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS13649; 2013-003884-71; U1111-1148-2987 (Other: UTN)
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2021-07-23 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alemtuzumab (Experimental): All Participants who completed the study CAMMS03409 (extension study of CAMMS223 [NCT00050778], CAMMS323 [NCT00530348], or CAMMS324 [NCT00548405]) and received alemtuzumab within 48 months prior to enrollment were included in this LPS13649 study. Participants received alemtuzumab, intravenous infusion of 12 milligram per day (mg/day) for 3 consecutive days, at the study investigators' discretion; and at least 12 months after the prior treatment course in the current study (LPS13649).
  Interventions: Drug: alemtuzumab GZ402673

INTERVENTIONS:
Drug: alemtuzumab GZ402673 — Pharmaceutical form:concentrate for solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objective:

To evaluate long-term safety of alemtuzumab.

Secondary Objectives:

* To evaluate long term efficacy of alemtuzumab.
* To evaluate the safety profile of participants who received other Disease Modifying Treatment (DMT) following alemtuzumab treatment.
* To evaluate participant-reported Quality of Life (QoL) outcomes and health resource utilization of participant who received alemtuzumab.
* To evaluate as needed re-treatment with alemtuzumab and other DMTs.

DETAILED DESCRIPTION:
The total duration per participants was up to 5.6 years.

As per Study Investigator discretion, participants can be treated with additional courses of alemtuzumab or any commercialized DMTs.

All participants who completed CAMMS03409 were allowed into the study, which might include specific vulnerable populations. If the investigator decided to treat a participant with a course of alemtuzumab, appropriate cautionary measures were applied as indicated in the approved labelling, or, in ex-European Union countries where Lemtrada was not approved, according to the investigator's brochure.

ELIGIBILITY:
Inclusion criteria:

Participant had completed at least 48 months of the Extension Study CAMMS03409. Signed written informed consent form.

Exclusion criteria:

Participant participating in another investigational interventional study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1062 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (131):
- United States (52):
  - Investigational Site Number 1086, Cullman, Alabama
  - Investigational Site Number 1031, Phoenix, Arizona
  - Investigational Site Number 1171, Phoenix, Arizona
  - Investigational Site Number 1090, Tucson, Arizona
  - Investigational Site Number 1040, Berkeley, California
  - Investigational Site Number 1152, Fullerton, California
  - Investigational Site Number 1093, Pasadena, California
  - Investigational Site Number 1027, Fort Collins, Colorado
  - Investigational Site Number 1078, Jacksonville, Florida
  - Investigational Site Number 1059, Maitland, Florida
  - Investigational Site Number 1173, Sarasota, Florida
  - Investigational Site Number 1034, Sunrise, Florida
  - Investigational Site Number 1005, Tampa, Florida
  - Investigational Site Number 1049, Tampa, Florida
  - Investigational Site Number 1008, Northbrook, Illinois
  - Investigational Site Number 1001, Fort Wayne, Indiana
  - Investigational Site Number 1024, Indianapolis, Indiana
  - Investigational Site Number 1017, Des Moines, Iowa
  - Investigational Site Number 1022, Kansas City, Kansas
  - Investigational Site Number 1083, Lenexa, Kansas
  - Investigational Site Number 1039, Lexington, Kentucky
  - Investigational Site Number 1021, Louisville, Kentucky
  - Investigational Site Number 1061, Wellesley, Massachusetts
  - Investigational Site Number 1028, Worcester, Massachusetts
  - Investigational Site Number 1025, Ann Arbor, Michigan
  - Investigational Site Number 1020, Detroit, Michigan
  - Investigational Site Number 1054, Traverse City, Michigan
  - Investigational Site Number 1084, Kansas City, Missouri
  - Investigational Site Number 1092, St Louis, Missouri
  - Investigational Site Number 1073, Teaneck, New Jersey
  - Investigational Site Number 1014, Albuquerque, New Mexico
  - Investigational Site Number 1081, Mineola, New York
  - Investigational Site Number 1026, New York, New York
  - Investigational Site Number 1160, Patchogue, New York
  - Investigational Site Number 1015, Rochester, New York
  - Investigational Site Number 1053, Syracuse, New York
  - Investigational Site Number 1095, Chapel Hill, North Carolina
  - Investigational Site Number 1082, Winston-Salem, North Carolina
  - Investigational Site Number 1035, Cleveland, Ohio
  - Investigational Site Number 1058, Uniontown, Ohio
  - Investigational Site Number 1067, Oklahoma City, Oklahoma
  - Investigational Site Number 1097, Allentown, Pennsylvania
  - Investigational Site Number 1057, Providence, Rhode Island
  - Investigational Site Number 1163, Cordova, Tennessee
  - Investigational Site Number 1055, Franklin, Tennessee
  - Investigational Site Number 1009, Knoxville, Tennessee
  - Investigational Site Number 1042, Nashville, Tennessee
  - Investigational Site Number 1018, Houston, Texas
  - Investigational Site Number 1002, Round Rock, Texas
  - Investigational Site Number 1046, San Antonio, Texas
  - Investigational Site Number 1037, Vienna, Virginia
  - Investigational Site Number 1068, Seattle, Washington
- Investigational Site Number 03208, CABA, Argentina
- Australia (9):
  - Investigational Site Number 2013, Auchenflower
  - Investigational Site Number 2001, Heidelberg
  - Investigational Site Number 2011, Hobart
  - Investigational Site Number 2012, Kogarah
  - Investigational Site Number 2003, Melbourne
  - Investigational Site Number 2002, Parkville
  - Investigational Site Number 2005, Southport
  - Investigational Site Number 2009, Sydney
  - Investigational Site Number 2006, Westmead
- Belgium (3):
  - Investigational Site Number 5005, Brussels
  - Investigational Site Number 5004, Esneux
  - Investigational Site Number 5001, Leuven
- Brazil (4):
  - Investigational Site Number 3006, Porto Alegre
  - Investigational Site Number 3002, Recife
  - Investigational Site Number 3001, São Paulo
  - Investigational Site Number 3003, São Paulo
- Canada (7):
  - Investigational Site Number 1102, Calgary
  - Investigational Site Number 1105, Gatineau
  - Investigational Site Number 1104, Greenfield Park
  - Investigational Site Number 1109, Kingston
  - Investigational Site Number 1110, London
  - Investigational Site Number 1101, Ottawa
  - Investigational Site Number 1106, Vancouver
- Czechia (4):
  - Investigational Site Number 4803, Brno
  - Investigational Site Number 4804, Hradec Králové
  - Investigational Site Number 4801, Prague
  - Investigational Site Number 4802, Teplice
- Denmark (2):
  - Investigational Site Number 5302, Aarhus N
  - Investigational Site Number 5301, København Ø
- Germany (9):
  - Investigational Site Number 4602, Berlin
  - Investigational Site Number 4607, Dresden
  - Investigational Site Number 4634, Frankfurt am Main
  - Investigational Site Number 4622, Hamburg
  - Investigational Site Number 4605, Hanover
  - Investigational Site Number 4609, Hennigsdorf
  - Investigational Site Number 4608, München
  - Investigational Site Number 4610, Rostock
  - Investigational Site Number 4613, Wermsdorf
- Israel (2):
  - Investigational Site Number 5501, Ramat Gan
  - Investigational Site Number 5505, Tel Aviv
- Italy (4):
  - Investigational Site Number 4112, Cagliari
  - Investigational Site Number 4102, Gallarate (VA)
  - Investigational Site Number 4106, Orbassano (TO)
  - Investigational Site Number 4110, Roma
- Mexico (2):
  - Investigational Site Number 3105, Chihuahua City
  - Investigational Site Number 3102, México
- Investigational Site Number 4202, Sittard-Geleen, Netherlands
- Poland (5):
  - Investigational Site Number 4902, Krakow
  - Investigational Site Number 4901, Lodz
  - Investigational Site Number 4903, Lublin
  - Investigational Site Number 4904, Poznan
  - Investigational Site Number 4905, Warsaw
- Russia (11):
  - Investigational Site Number 6009, Kazan'
  - Investigational Site Number 6001, Moscow
  - Investigational Site Number 6005, Moscow
  - Investigational Site Number 6003, Moscow
  - Investigational Site Number 6006, Nizhny Novgorod
  - Investigational Site Number 6010, Pyatigorsk
  - Investigational Site Number 6002, Saint Petersburg
  - Investigational Site Number 6004, Saint Petersburg
  - Investigational Site Number 6008, Saint Petersburg
  - Investigational Site Number 6013, Samara
  - Investigational Site Number 6016, Ufa
- Spain (4):
  - Investigational Site Number 4301, Barcelona
  - Investigational Site Number 4303, Madrid
  - Investigational Site Number 4305, Málaga
  - Investigational Site Number 4304, Seville
- Sweden (2):
  - Investigational Site Number 4701, Gothenburg
  - Investigational Site Number 4702, Umeå
- Ukraine (3):
  - Investigational Site Number 6102, Kharkiv
  - Investigational Site Number 6104, Kiev
  - Investigational Site Number 6103, Lviv
- United Kingdom (6):
  - Investigational Site Number 4004, Bristol
  - Investigational Site Number 4001, Cambridge
  - Investigational Site Number 4005, Cardiff
  - Investigational Site Number 4006, London
  - Investigational Site Number 4008, Salford
  - Investigational Site Number 4007, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Ziemssen T, Bass AD, Van Wijmeersch B, Eichau S, Richter S, Hoffmann F, Armstrong NM, Chirieac M, Cunha-Santos J, Singer BA. Long-term efficacy and safety of alemtuzumab in participants with highly active MS: TOPAZ clinical trial and interim analysis of TREAT-MS real-world study. Ther Adv Neurol Disord. 2025 Feb 10;18:17562864241306575. doi: 10.1177/17562864241306575. eCollection 2025. PMID 39935588
- [Derived] Coles AJ, Achiron A, Traboulsee A, Singer BA, Pozzilli C, Oreja-Guevara C, Giovannoni G, Comi G, Freedman MS, Ziemssen T, Shiota D, Rawlings AM, Wong AT, Chirieac M, Montalban X. Safety and efficacy with alemtuzumab over 13 years in relapsing-remitting multiple sclerosis: final results from the open-label TOPAZ study. Ther Adv Neurol Disord. 2023 Sep 21;16:17562864231194823. doi: 10.1177/17562864231194823. eCollection 2023. PMID 37745914
- [Derived] Coles AJ, Jones JL, Vermersch P, Traboulsee A, Bass AD, Boster A, Chan A, Comi G, Fernandez O, Giovannoni G, Kubala Havrdova E, LaGanke C, Montalban X, Oreja-Guevara C, Piehl F, Wiendl H, Ziemssen T. Autoimmunity and long-term safety and efficacy of alemtuzumab for multiple sclerosis: Benefit/risk following review of trial and post-marketing data. Mult Scler. 2022 Apr;28(5):842-846. doi: 10.1177/13524585211061335. Epub 2021 Dec 9. PMID 34882037
- [Derived] Kuhle J, Daizadeh N, Benkert P, Maceski A, Barro C, Michalak Z, Sormani MP, Godin J, Shankara S, Samad TA, Jacobs A, Chung L, Rӧsch N, Kaiser C, Mitchell CP, Leppert D, Havari E, Kappos L. Sustained reduction of serum neurofilament light chain over 7 years by alemtuzumab in early relapsing-remitting MS. Mult Scler. 2022 Apr;28(4):573-582. doi: 10.1177/13524585211032348. Epub 2021 Aug 11. PMID 34378446
- [Derived] Bass AD, Arroyo R, Boster AL, Boyko AN, Eichau S, Ionete C, Limmroth V, Navas C, Pelletier D, Pozzilli C, Ravenscroft J, Sousa L, Tintore M, Uitdehaag BMJ, Baker DP, Daizadeh N, Choudhry Z, Rog D; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ investigators. Alemtuzumab outcomes by age: Post hoc analysis from the randomized CARE-MS studies over 8 years. Mult Scler Relat Disord. 2021 Apr;49:102717. doi: 10.1016/j.msard.2020.102717. Epub 2020 Dec 24. PMID 33476880
- [Derived] Ziemssen T, Bass AD, Berkovich R, Comi G, Eichau S, Hobart J, Hunter SF, LaGanke C, Limmroth V, Pelletier D, Pozzilli C, Schippling S, Sousa L, Traboulsee A, Uitdehaag BMJ, Van Wijmeersch B, Choudhry Z, Daizadeh N, Singer BA; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ investigators. Efficacy and Safety of Alemtuzumab Through 9 Years of Follow-up in Patients with Highly Active Disease: Post Hoc Analysis of CARE-MS I and II Patients in the TOPAZ Extension Study. CNS Drugs. 2020 Sep;34(9):973-988. doi: 10.1007/s40263-020-00749-x. PMID 32710396
- [Derived] Steingo B, Al Malik Y, Bass AD, Berkovich R, Carraro M, Fernandez O, Ionete C, Massacesi L, Meuth SG, Mitsikostas DD, Pardo G, Simm RF, Traboulsee A, Choudhry Z, Daizadeh N, Compston DAS; CAMMS223, CAMMS03409, and TOPAZ Investigators. Long-term efficacy and safety of alemtuzumab in patients with RRMS: 12-year follow-up of CAMMS223. J Neurol. 2020 Nov;267(11):3343-3353. doi: 10.1007/s00415-020-09983-1. Epub 2020 Jun 24. PMID 32583052
- [Derived] Comi G, Alroughani R, Boster AL, Bass AD, Berkovich R, Fernandez O, Kim HJ, Limmroth V, Lycke J, Macdonell RA, Sharrack B, Singer BA, Vermersch P, Wiendl H, Ziemssen T, Jacobs A, Daizadeh N, Rodriguez CE, Traboulsee A; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ Investigators. Efficacy of alemtuzumab in relapsing-remitting MS patients who received additional courses after the initial two courses: Pooled analysis of the CARE-MS, extension, and TOPAZ studies. Mult Scler. 2020 Dec;26(14):1866-1876. doi: 10.1177/1352458519888610. Epub 2019 Nov 25. PMID 31762387
- [Derived] Okai AF, Amezcua L, Berkovich RR, Chinea AR, Edwards KR, Steingo B, Walker A, Jacobs AK, Daizadeh N, Williams MJ; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ Investigators. Efficacy and Safety of Alemtuzumab in Patients of African Descent with Relapsing-Remitting Multiple Sclerosis: 8-Year Follow-up of CARE-MS I and II (TOPAZ Study). Neurol Ther. 2019 Dec;8(2):367-381. doi: 10.1007/s40120-019-00159-2. Epub 2019 Oct 25. PMID 31654272

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 142 study centers in 21 countries. A total of 1062 participants were screened between 7 January 2015 and 28 June 2016 and were enrolled in this current study (LPS13649 [TOPAZ]).
Pre-assignment Details: Subgroup analysis ([Delayed Alemtuzumab Treatment[DAT] & Immediate Alemtuzumab Treatment[IAT]subgroup) was performed only for outcome measures and safety analysis. Participants who rolled over from CAMMS223(NCT00050778) to CAMMS03409 (NCT00930553),then subsequently enrolled and took 24 mg alemtuzumab in CAMMS324 (NCT00548405) study, were not considered as part of DAT or IAT subgroup & included in overall group only. Participant flow and Baseline analysis was performed on overall population only.
Period: Overall Study
Arm/Group | Alemtuzumab
Started | 1062
Completed | 592
Not Completed | 470
Not completed — Adverse Event | 11
Not completed — Poor compliance to protocol | 3
Not completed — Lost to Follow-up | 30
Not completed — Due to Coronavirus Disease (Covid-19) | 300
Not completed — Other | 126

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- Alemtuzumab: All Participants who completed the study CAMMS03409 (extension study of CAMMS223 [NCT00050778], CAMMS323 [NCT00530348], or CAMMS324 [NCT00548405]) and received alemtuzumab within 48 months prior to enrollment were included in this LPS13649 study. Participants received alemtuzumab, intravenous infusion of 12 mg/day for 3 consecutive days, at the study investigators' discretion; and at least 12 months after the prior treatment course in the current study (LPS13649).
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1062
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 686
  Male | 376
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 988
  Black or African American | 34
  Asian | 5
  American Indian or Alaska native | 6
  Other | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) was any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily had to have causal relationship with treatment. TEAEs were defined as AEs that developed/worsened during the 'treatment period (time from Baseline until the end of the study LPS13649 [i.e. up to a maximum of 5.6 years]). Serious adverse events (SAEs) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: From Baseline until the end of the study (up to a maximum duration of 5.6 years)
Population: Analysis was performed on safety analysis set that included all participants who signed the informed consent form (ICF). As pre-specified, data collection and analysis for this outcome measure was done on the overall population along with 2 subgroups (DAT and IAT).
Measure: Count of Participants; unit: Participants
Groups:
- Delayed Alemtuzumab Treatment (DAT): Participants from the subcutaneous interferon beta-1a (SC IFNB1a) treatment arms of studies CAMMS323 and CAMMS324, who received their initial 2 treatment courses of alemtuzumab during the CAMMS03409 extension study were included in the DAT subgroup of the current study (LPS13649). Participants received alemtuzumab intravenous infusion of 12 mg/day for 3 consecutive days, at the study investigators' discretion; and at least 12 months after the prior treatment course in the current study (LPS13649).
- Initial Alemtuzumab Treatment (IAT): Participants from the 12 mg/day alemtuzumab treatment arms of the studies CAMMS323 and CAMMS324 (who were subsequently enrolled in CAMMS03409 extension study and then entered in this study LPS13649) were included in the IAT subgroup of the current study (LPS13649). Participants received alemtuzumab intravenous infusion of 12 mg/day for 3 consecutive days, at the study investigators' discretion; and at least 12 months after the prior treatment course in the current study (LPS13649).
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 241 | 598 | 1062
Participants
  Any TEAE | 204 | 500 | 879
  Any TESAE | 55 | 133 | 237
  Any TEAE leading to death | 0 | 10 | 11
  Any TEAE leading to permanent treatment discontinuation | 0 | 2 | 2

2. Primary Outcome: Number of Participants With Infusion-Associated Reactions (IAR)
Description: Infusion-associated reactions (IAR) was defined as any adverse event occurring during and within 24 hours of alemtuzumab infusion.
Time Frame: Within 24 hours of any alemtuzumab infusion
Population: Analysis was performed on re-treated population that included all participants who had signed the ICF and who had received study drug in the current study LPS13649. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. As pre-specified, data collection and analysis for this outcome measure was done on the overall population along with 2 subgroups (DAT and IAT).
Measure: Count of Participants; unit: Participants
Groups:
- Delayed Alemtuzumab Treatment (DAT): Participants from the SC IFNB1a treatment arms of studies CAMMS323 and CAMMS324, who received their initial 2 treatment courses of alemtuzumab during the CAMMS03409 extension study were included in the DAT subgroup of the current study (LPS13649). Participants received alemtuzumab intravenous infusion of 12 mg/day for 3 consecutive days, at the study investigators' discretion; and at least 12 months after the prior treatment course in the current study (LPS13649).
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 83 | 164 | 294
Participants | 48 | 89 | 164

3. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)
Description: Adverse events of special interest included the following: hypersensitivity or anaphylaxis; pregnancy of a woman entered in the study; symptomatic overdose (serious or non-serious) with investigational medicinal Product (IMP); increase in alanine transaminase (ALT); autoimmune mediated conditions; hemophagocytic lymphohistiocytosis; progressive multifocal leukoencephalopathy; temporally associated AEs; serious infections; malignancy; and pneumonitis.
Time Frame: From Baseline until the end of the study (up to a maximum duration of 5.6 years)
Population: Analysis was performed on safety population. As pre-specified, data collection and analysis for this outcome measure was done on the overall population along with 2 subgroups (DAT and IAT).
Measure: Count of Participants; unit: Participants
Groups:
- Alemtuzumab: All Participants who completed the study CAMMS03409 (extension study of CAMMS223 [NCT00050778], CAMMS323 [NCT00530348], and CAMMS324 [NCT00548405]) and received alemtuzumab within 48 months prior to enrollment were included in this LPS13649 study. Participants received alemtuzumab, intravenous infusion of 12 mg/day for 3 consecutive days, at the study investigators' discretion; and at least 12 months after the prior treatment course in the current study (LPS13649).
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 241 | 598 | 1062
Participants
  Hypersensitivity or anaphylaxis | 12 | 25 | 44
  Pregnancy of a woman entered in the study | 17 | 42 | 70
  Symptomatic overdose (serious or non-serious) with IMP | 0 | 0 | 0
  Increase in ALT | 0 | 0 | 1
  Autoimmune mediated conditions | 27 | 66 | 100
  Hemophagocytic lymphohistiocytosis | 0 | 0 | 0
  Progressive multifocal leukoencephalopathy | 0 | 0 | 0
  Temporally associated AEs | 2 | 4 | 9
  Serious infections | 10 | 35 | 60
  Malignancy | 6 | 15 | 27
  Pneumonitis | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities
Description: Criteria for potentially clinically significant laboratory abnormalities included:
  * Hemoglobin (Hb): less than or equal to (<=)115 grams per liter (g/L)(Male [M]), <= 95 g/L (Female[ F]); greater than or equal to (>=)185 g/L (M), >= 165 g/L (F); Decrease From Baseline (DFB) >= 20 g/L.
  * Hematocrit: <= 0.37 volume/volume (v/v) (M); <= 0.32 v/v (F); >= 0.55 v/v (M); >= 0.5 v/v (F).
  * Red Blood Cells (RBCs): >=6 *10^12/L.
  * Platelets: <100 *10^9/L; >=700 *10^9/L. As pre-specified, data collection and analysis for this outcome measure was done on the overall population along with 2 subgroups (DAT and IAT).
Time Frame: From Baseline until the end of the study (up to a maximum duration of 5.6 years)
Population: Analysis was performed on all participants who had signed the ICF; and received study drug in the TOPAZ study; or in studies CAMMS223,CAMMS323,CAMMS324 or CAMMS03409, and did not complete 48 months of follow-up at the screening visit in the TOPAZ study. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Groups:
- Alemtuzumab (Overall): All Participants who completed the study CAMMS03409 (extension study of CAMMS223 [NCT00050778], CAMMS323 [NCT00530348], or CAMMS324 [NCT00548405]) and received alemtuzumab within 48 months prior to enrollment were included in this LPS13649 study. Participants received alemtuzumab, intravenous infusion of 12 mg/day for 3 consecutive days, at the study investigators' discretion; and at least 12 months after the prior treatment course in the current study (LPS13649).
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab (Overall)
Number analyzed (Participants) | 214 | 316 | 619
Participants
  Hb:<=115 g/L, <=95 g/L | 11 | 28 | 43
  Hb: >=185 g/L, >=165 g/L | 2 | 6 | 12
  Hb: DFB >=20 g/L: number analyzed (Participants) | 206 | 293 | 580
  Hb: DFB >=20 g/L | 32 | 50 | 98
  Hematocrit: <= 0.37 v/v; <=0.32 v/v: number analyzed (Participants) | 213 | 315 | 617
  Hematocrit: <= 0.37 v/v; <=0.32 v/v | 20 | 42 | 70
  Hematocrit: >=0.55 v/v; >=0.5 v/v: number analyzed (Participants) | 213 | 315 | 617
  Hematocrit: >=0.55 v/v; >=0.5 v/v | 6 | 14 | 26
  RBCs: >=6 *10^12/L: number analyzed (Participants) | 214 | 315 | 618
  RBCs: >=6 *10^12/L | 8 | 7 | 21
  Platelets: <100 *10^9/L: number analyzed (Participants) | 212 | 314 | 615
  Platelets: <100 *10^9/L | 5 | 16 | 25
  Platelets: >=700 *10^9/L: number analyzed (Participants) | 212 | 314 | 615
  Platelets: >=700 *10^9/L | 1 | 0 | 1

5. Secondary Outcome: Annualized Relapse Rate
Description: Relapse was defined as new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination. Annualized relapse rate was obtained from the total number of confirmed relapses that occurred during the treatment follow up time of all participants divided by the total years of follow-up for all participants. The annualized relapse rate was estimated using a negative binomial model with robust variance estimation.
Time Frame: Up to a maximum duration of 5.6 years
Population: Analysis was performed on efficacy population which included all enrolled participants who had received study drug in studies CAMMS223, CAMMS323, CAMMS324 or CAMMS03409. As pre-specified, data collection and analysis for this outcome measure was done only on the 2 subgroups (DAT and IAT).
Measure: Number (95% Confidence Interval); unit: relapses per participant per year
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
relapses per participant per year | 0.1994 [0.1710 to 0.2325] | 0.1608 [0.1418 to 0.1823]

6. Secondary Outcome: Proportion of Participants Who Were Relapse Free
Description: Relapse was defined as new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination. The proportion of participants who were relapse free (without event) were estimated using the Kaplan-Meier method.
Time Frame: Up to a maximum duration of 5.6 years
Population: Analysis was performed on efficacy population. As pre-specified, data collection and analysis for this outcome measure was done only on the 2 subgroups (DAT and IAT).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
proportion of participants | 29.59 [23.73 to 35.65] | 36.86 [32.96 to 40.76]

7. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score at Month 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in participants with multiple sclerosis (MS). It consists of 8 ordinal rating scales assessing seven functional systems (pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral, and other). EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicated worst outcomes.
Time Frame: Baseline (Month 0 of LPS13649), Month 6, 12, 18, 24, 30, 36, 42, 48, 54 and 60
Population: Analysis was performed on efficacy population. Here, 'Number analyzed' = participants with available data for each specified category. As pre-specified, data collection and analysis for this outcome measure was done only on the 2 subgroups (DAT and IAT).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
score on a scale
  Month 6: number analyzed (Participants) | 237 | 583
  Month 6 | 0.21 (0.092) | 0.03 (0.065)
  Month 12: number analyzed (Participants) | 234 | 580
  Month 12 | 0.27 (0.093) | 0.08 (0.065)
  Month 18: number analyzed (Participants) | 226 | 562
  Month 18 | 0.29 (0.096) | 0.10 (0.067)
  Month 24: number analyzed (Participants) | 227 | 559
  Month 24 | 0.28 (0.102) | 0.15 (0.070)
  Month 30: number analyzed (Participants) | 225 | 547
  Month 30 | 0.34 (0.102) | 0.16 (0.071)
  Month 36: number analyzed (Participants) | 219 | 545
  Month 36 | 0.38 (0.103) | 0.18 (0.071)
  Month 42: number analyzed (Participants) | 217 | 515
  Month 42 | 0.37 (0.103) | 0.24 (0.071)
  Month 48: number analyzed (Participants) | 204 | 468
  Month 48 | 0.46 (0.104) | 0.27 (0.072)
  Month 54: number analyzed (Participants) | 168 | 346
  Month 54 | 0.51 (0.106) | 0.30 (0.074)
  Month 60: number analyzed (Participants) | 55 | 125
  Month 60 | 0.43 (0.129) | 0.32 (0.088)

8. Secondary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Number of Gadolinium Enhancing (Gd-enhancing) Lesions Per MRI Scan
Description: Number of Gd-enhancing lesions per scan was defined as the total number of Gd-enhancing lesions that occurred during the treatment period divided by the total number of scans performed during the treatment period. The adjusted cumulative count of lesions was estimated by a repeated negative binomial regression with generalized estimating equation (GEE) adjusted for analysis groups and geographic region as covariates.
Time Frame: Up to a maximum duration of 5.6 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
lesions per scan | 1.307 [0.880 to 1.941] | 1.558 [1.153 to 2.105]

9. Secondary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Number of New or Enlarged T2 Lesions Per MRI Scan
Description: Number of new or enlarged T2 lesions per scan was defined as the total number of new or enlarged T2 lesion that occurred during treatment period divided by the total number of scans performed during treatment period. The adjusted cumulative count of lesions was estimated by a repeated negative binomial regression with GEE adjusted for analysis groups and geographic region as covariates.
Time Frame: Up to a maximum duration of 5.6 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
lesions per scan | 8.033 [6.001 to 10.753] | 9.564 [7.656 to 11.946]

10. Secondary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Number of New T1 (and New Hypointense T1) Lesions Per MRI Scan
Description: Number of new T1 lesions per scan was defined as the total number of new T1 lesion (and New Hypointense T1) that occurred during treatment period divided by the total number of scans performed during treatment period.The adjusted cumulative count of lesions was estimated by a repeated negative binomial regression with GEE adjusted for analysis groups and geographic region as covariates.
Time Frame: Up to a maximum duration of 5.6 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
lesions per scan | 1.719 [1.141 to 2.589] | 1.908 [1.386 to 2.628]

11. Secondary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Percent Change From Baseline in Volume of T1 Lesions at Months 12, 24, 36, 48, and 60
Description: The total lesion volume (T1 lesions) was measured by MRI scan.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: Analysis was preformed on efficacy population. Here, 'Number analyzed' = participants with available data for each specified category. As pre-specified, data collection and analysis for this outcome measure was done only on the 2 subgroups (DAT and IAT).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
percent change
  Month 12: number analyzed (Participants) | 203 | 501
  Month 12 | 141.71 (449.79) | 64.73 (241.92)
  Month 24: number analyzed (Participants) | 202 | 489
  Month 24 | 130.73 (398.65) | 67.48 (262.64)
  Month 36: number analyzed (Participants) | 194 | 478
  Month 36 | 145.57 (404.35) | 104.41 (524.62)
  Month 48: number analyzed (Participants) | 185 | 421
  Month 48 | 163.30 (461.38) | 76.90 (312.05)
  Month 60: number analyzed (Participants) | 60 | 116
  Month 60 | 202.47 (499.46) | 93.61 (260.51)

12. Secondary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Percent Change From Baseline in Volume of T2 Lesions at Months 12, 24, 36, 48, and 60
Description: The total lesion volume (T2 lesions) was measured by MRI scan.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
percent change
  Month 12: number analyzed (Participants) | 226 | 558
  Month 12 | 21.44 (132.04) | 9.09 (62.52)
  Month 24: number analyzed (Participants) | 224 | 542
  Month 24 | 17.53 (76.73) | 13.89 (62.45)
  Month 36: number analyzed (Participants) | 216 | 529
  Month 36 | 24.24 (94.85) | 22.02 (111.95)
  Month 48: number analyzed (Participants) | 204 | 462
  Month 48 | 21.98 (80.06) | 19.46 (70.72)
  Month 60: number analyzed (Participants) | 67 | 128
  Month 60 | 32.03 (136.68) | 17.95 (75.47)

13. Secondary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Percent Change From Baseline in Brain Parenchymal Fraction (BPF) at Month 12, 24, 36, 48, and 60
Description: The brain parenchymal fraction was measured by MRI scan.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
percent change
  Month 12: number analyzed (Participants) | 221 | 549
  Month 12 | -1.65 (1.59) | -1.49 (1.55)
  Month 24: number analyzed (Participants) | 220 | 534
  Month 24 | -1.77 (1.56) | -1.68 (1.64)
  Month 36: number analyzed (Participants) | 215 | 524
  Month 36 | -1.92 (1.56) | -1.84 (1.71)
  Month 48: number analyzed (Participants) | 203 | 459
  Month 48 | -2.02 (1.58) | -2.07 (1.78)
  Month 60: number analyzed (Participants) | 66 | 129
  Month 60 | -2.11 (1.67) | -2.37 (1.65)

14. Secondary Outcome: Change From Baseline in Self-reported Quality of Life (QoL) as Assessed by the Medical Outcome Study (MOS) 36-Item Short-Form Health Survey (SF-36): Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores at Month 12, 24, 36, 48, and 60
Description: The MOS SF-36 is an extensively validated and widely used measure of QoL that assesses participants' perceptions of health status and its impact on their lives. It consisted of 36 items organized into 8 scales (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health). Two summary measures of physical and mental health, the PCS and MCS, respectively, were derived from scale aggregates, and were reported in this outcome measure. The score range for each of these 2 summary scores was from 0 (worst) to 100 (best), higher scores indicated better QoL.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
score on a scale
  PCS: Month 12: number analyzed (Participants) | 228 | 559
  PCS: Month 12 | 0.54 (9.38) | 0.88 (8.72)
  PCS: Month 24: number analyzed (Participants) | 216 | 545
  PCS: Month 24 | 0.20 (9.25) | 0.59 (9.10)
  PCS: Month 36: number analyzed (Participants) | 212 | 534
  PCS: Month 36 | 0.08 (9.88) | 1.12 (9.18)
  PCS: Month 48: number analyzed (Participants) | 199 | 466
  PCS: Month 48 | -0.52 (10.15) | 0.68 (9.57)
  PCS: Month 60: number analyzed (Participants) | 80 | 176
  PCS: Month 60 | -0.23 (8.85) | 1.28 (8.88)
  MCS: Month 12: number analyzed (Participants) | 228 | 559
  MCS: Month 12 | 2.21 (12.29) | 0.89 (11.24)
  MCS: Month 24: number analyzed (Participants) | 216 | 545
  MCS: Month 24 | 1.21 (12.23) | 1.11 (11.93)
  MCS: Month 36: number analyzed (Participants) | 212 | 534
  MCS: Month 36 | 1.55 (12.23) | 0.94 (11.88)
  MCS: Month 48: number analyzed (Participants) | 199 | 466
  MCS: Month 48 | 1.14 (12.93) | 0.35 (12.38)
  MCS: Month 60: number analyzed (Participants) | 80 | 176
  MCS: Month 60 | 0.94 (14.01) | 0.45 (11.39)

15. Secondary Outcome: Change From Baseline in Functional Assessment of Multiple Sclerosis (FAMS) Score at Month 12, 24, 36, 48, and 60
Description: The FAMS is a self-reported multidimensional index comprising a total of 58 items on 7 subscales: mobility (7 items); symptoms (7 items); emotional well-being (7 items); general contentment (7 items); thinking and fatigue (9 items); family/social well-being (7 items); and additional concerns (14 items, these are not scored). Each item (except those for "additional concerns") was rated on a 5-point scale of 0 (lower quality of life) to 4 (higher quality of life). Total FAMS score was the sum of 44 scored items, which ranged from 0 (poor) to 176 (best), with higher numbers reflecting a higher quality of life.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
score on a scale
  Month 12: number analyzed (Participants) | 230 | 573
  Month 12 | 1.05 (29.68) | 2.83 (27.07)
  Month 24: number analyzed (Participants) | 222 | 551
  Month 24 | -0.45 (30.30) | 2.73 (28.62)
  Month 36: number analyzed (Participants) | 214 | 532
  Month 36 | 0.82 (30.52) | 2.70 (28.94)
  Month 48: number analyzed (Participants) | 202 | 472
  Month 48 | -3.73 (31.46) | 1.16 (29.38)
  Month 60: number analyzed (Participants) | 81 | 181
  Month 60 | -0.36 (31.25) | 2.74 (26.61)

16. Secondary Outcome: Change From Baseline in European Quality of Life -5 Dimension (EQ-5D) Score: Utility Scores at Month 12, 24, 36, 48, and 60
Description: The EQ-5D is a generic, standardized instrument that provides a simple, descriptive profile and a single index value for health status used in the clinical and economic evaluation of health care as well as in population health surveys. The EQ-5D comprises 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension measured on 3 levels: some, moderate, and extreme problems. The 5 dimensional 3-level systems was converted into single index utility score ranges from 0 to 100, where 100=best health state; and 0=worst health state; higher scores indicated better outcome.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
score on a scale
  Month 12: number analyzed (Participants) | 231 | 571
  Month 12 | -0.01 (0.26) | -0.01 (0.26)
  Month 24: number analyzed (Participants) | 225 | 550
  Month 24 | -0.02 (0.28) | -0.01 (0.26)
  Month 36: number analyzed (Participants) | 218 | 530
  Month 36 | -0.04 (0.27) | -0.00 (0.26)
  Month 48: number analyzed (Participants) | 207 | 469
  Month 48 | -0.03 (0.27) | -0.03 (0.27)
  Month 60: number analyzed (Participants) | 83 | 184
  Month 60 | -0.03 (0.29) | -0.03 (0.25)

17. Secondary Outcome: Change From Baseline in EQ-5D Visual Analogue Scale (VAS) Scores at Month 12, 24, 36, 48, and 60
Description: EQ-5D VAS was used to record a participant's rating for his/her current health-related quality of life state and captured on a vertical VAS (0 to 100), where 0=worst imaginable health state to 100=best imaginable health state, and higher score indicated better outcome.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT)
Number analyzed (Participants) | 241 | 598
score on a scale
  Month 12: number analyzed (Participants) | 232 | 560
  Month 12 | -2.09 (25.11) | -1.05 (24.57)
  Month 24: number analyzed (Participants) | 225 | 545
  Month 24 | -1.57 (26.69) | -0.39 (21.44)
  Month 36: number analyzed (Participants) | 217 | 527
  Month 36 | 0.10 (22.61) | 1.42 (20.64)
  Month 48: number analyzed (Participants) | 199 | 466
  Month 48 | -1.08 (23.66) | -0.85 (23.94)
  Month 60: number analyzed (Participants) | 82 | 177
  Month 60 | -3.26 (27.04) | -0.77 (26.26)

18. Secondary Outcome: Modified Healthcare Resource Utilization Questionnaire (HRUQ): Number of Participants Who Reported Change in Employment Situation, Availing of Sick Leaves, Admissions and Stays in Hospital, Rehabilitation Centers or Nursing Homes Due to Multiple Sclerosis
Description: Participants use of healthcare resources, non-medical resources, and informal care as well as their work capacity was assessed at scheduled study visits using a modified questionnaire (HRUQ) designed to evaluate the economic impact of MS. Questionnaire addresses the following content areas: employment situation and changes in employment situation due to MS;sick leaves,admissions and stays in hospital, rehabilitation centers, or nursing homes; typical MS-related investments (eg, stair and bed lift, ramps,rails) and devices (eg,walking aids,wheelchairs); assistance by community or social services (e.g. home nurse, transportation), or help from family or friends. Each question requires a binary answer (yes/no). Number of participants who reported "Yes" as an answer to "employment situation change; had sick leaves; had hospital admission; had spent time in rehabilitation center and had spent time in a nursing home or a similar institution" questions were reported in this outcome measure.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: Analysis was performed on efficacy population. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants with available data for each specified category. As pre-specified, data collection and analysis for this outcome measure was done on the overall population along with 2 subgroups (DAT and IAT).
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 231 | 573 | 1020
Participants
  Employment situation change: Month 0: number analyzed (Participants) | 84 | 224 | 381
  Employment situation change: Month 0 | 3 | 7 | 12
  Employment situation change: Month 12: number analyzed (Participants) | 230 | 573 | 1014
  Employment situation change: Month 12 | 11 | 25 | 44
  Employment situation change: Month 24: number analyzed (Participants) | 220 | 537 | 960
  Employment situation change: Month 24 | 14 | 19 | 40
  Employment situation change: Month 36: number analyzed (Participants) | 217 | 518 | 929
  Employment situation change: Month 36 | 12 | 26 | 44
  Employment situation change: Month 48: number analyzed (Participants) | 200 | 467 | 850
  Employment situation change: Month 48 | 4 | 24 | 38
  Employment situation change: Month 60: number analyzed (Participants) | 81 | 182 | 367
  Employment situation change: Month 60 | 3 | 8 | 14
  Had sick leaves: Month 0: number analyzed (Participants) | 57 | 157 | 265
  Had sick leaves: Month 0 | 6 | 14 | 21
  Had sick leaves: Month 12: number analyzed (Participants) | 127 | 373 | 642
  Had sick leaves: Month 12 | 19 | 45 | 77
  Had sick leaves: Month 24: number analyzed (Participants) | 148 | 360 | 645
  Had sick leaves: Month 24 | 23 | 42 | 80
  Had sick leaves: Month 36: number analyzed (Participants) | 145 | 324 | 584
  Had sick leaves: Month 36 | 21 | 44 | 78
  Had sick leaves: Month 48: number analyzed (Participants) | 134 | 307 | 565
  Had sick leaves: Month 48 | 18 | 31 | 60
  Had sick leaves: Month 60: number analyzed (Participants) | 56 | 127 | 266
  Had sick leaves: Month 60 | 9 | 10 | 25
  Had hospital admission: Month 0: number analyzed (Participants) | 73 | 203 | 337
  Had hospital admission: Month 0 | 4 | 23 | 32
  Had hospital admission: Month 12: number analyzed (Participants) | 231 | 570 | 1018
  Had hospital admission: Month 12 | 28 | 59 | 109
  Had hospital admission: Month 24: number analyzed (Participants) | 223 | 544 | 974
  Had hospital admission: Month 24 | 26 | 53 | 95
  Had hospital admission: Month 36: number analyzed (Participants) | 218 | 522 | 938
  Had hospital admission: Month 36 | 27 | 58 | 106
  Had hospital admission: Month 48: number analyzed (Participants) | 202 | 471 | 859
  Had hospital admission: Month 48 | 20 | 51 | 89
  Had hospital admission: Month 60: number analyzed (Participants) | 81 | 184 | 374
  Had hospital admission: Month 60 | 12 | 11 | 28
  Had spent time in rehabilitation center: Month 0: number analyzed (Participants) | 74 | 200 | 334
  Had spent time in rehabilitation center: Month 0 | 0 | 6 | 8
  Had spent time in rehabilitation center: Month 12: number analyzed (Participants) | 230 | 573 | 1020
  Had spent time in rehabilitation center: Month 12 | 12 | 21 | 45
  Had spent time in rehabilitation center: Month 24: number analyzed (Participants) | 223 | 540 | 968
  Had spent time in rehabilitation center: Month 24 | 17 | 18 | 45
  Had spent time in rehabilitation center: Month 36: number analyzed (Participants) | 217 | 532 | 946
  Had spent time in rehabilitation center: Month 36 | 12 | 19 | 36
  Had spent time in rehabilitation center: Month 48: number analyzed (Participants) | 203 | 474 | 864
  Had spent time in rehabilitation center: Month 48 | 12 | 24 | 45
  Had spent time in rehabilitation center: Month 60: number analyzed (Participants) | 81 | 184 | 374
  Had spent time in rehabilitation center: Month 60 | 5 | 6 | 18
  Had spent time in a nursing home: Month 0: number analyzed (Participants) | 73 | 198 | 332
  Had spent time in a nursing home: Month 0 | 0 | 0 | 0
  Had spent time in a nursing home: Month 12: number analyzed (Participants) | 229 | 572 | 1019
  Had spent time in a nursing home: Month 12 | 0 | 5 | 8
  Had spent time in a nursing home: Month 24: number analyzed (Participants) | 222 | 545 | 972
  Had spent time in a nursing home: Month 24 | 3 | 4 | 7
  Had spent time in a nursing home: Month 36: number analyzed (Participants) | 218 | 523 | 938
  Had spent time in a nursing home: Month 36 | 3 | 3 | 8
  Had spent time in a nursing home: Month 48: number analyzed (Participants) | 202 | 472 | 860
  Had spent time in a nursing home: Month 48 | 4 | 4 | 11
  Had spent time in a nursing home: Month 60: number analyzed (Participants) | 81 | 184 | 369
  Had spent time in a nursing home: Month 60 | 0 | 4 | 6

19. Secondary Outcome: Modified HRUQ: Number of Participants Who Reported Other Changes/Changes in Lifestyle Due to Multiple Sclerosis
Description: Participants use of healthcare resources, non-medical resources, and informal care as well as their work capacity was assessed at scheduled study visits using a modified questionnaire (HRUQ) designed to evaluate the economic impact of MS.Questionnaire addresses following content areas: employment situation and changes in employment situation due to MS; admissions and stays in hospital, rehabilitation centers, or nursing homes; typical MS-related investments(e.g.stair and bed lift,ramps,rails) and devices(e.g.walking aids,wheelchairs);assistance by community or social services(e.g.home nurse, transportation), or help from family or friends. Each question requires a binary answer (yes/no). Number of participants who reported other changes/changes in lifestyle due to MS, i.e."Yes" as an answer to "had made changes to your house, apartment, car or did you require any special equipment or aids; assistance required; other assistance required" questions were reported in this outcome measure.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 231 | 573 | 1020
Participants
  Had made changes to your house, apartment, car: Month 0: number analyzed (Participants) | 75 | 202 | 339
  Had made changes to your house, apartment, car: Month 0 | 0 | 3 | 7
  Had made changes to your house, apartment, car: Month 12: number analyzed (Participants) | 231 | 571 | 1020
  Had made changes to your house, apartment, car: Month 12 | 11 | 21 | 42
  Had made changes to your house, apartment, car: Month 24: number analyzed (Participants) | 222 | 544 | 972
  Had made changes to your house, apartment, car: Month 24 | 10 | 25 | 47
  Had made changes to your house, apartment, car: Month 36: number analyzed (Participants) | 219 | 527 | 944
  Had made changes to your house, apartment, car: Month 36 | 16 | 15 | 45
  Had made changes to your house, apartment, car: Month 48: number analyzed (Participants) | 203 | 472 | 859
  Had made changes to your house, apartment, car: Month 48 | 10 | 25 | 42
  Had made changes to your house, apartment, car: Month 60: number analyzed (Participants) | 80 | 185 | 372
  Had made changes to your house, apartment, car: Month 60 | 5 | 3 | 12
  Had required assistance: Month 0: number analyzed (Participants) | 72 | 201 | 335
  Had required assistance: Month 0 | 4 | 10 | 24
  Had required assistance: Month 12: number analyzed (Participants) | 227 | 573 | 1015
  Had required assistance: Month 12 | 24 | 45 | 88
  Had required assistance: Month 24: number analyzed (Participants) | 221 | 535 | 962
  Had required assistance: Month 24 | 26 | 44 | 86
  Had required assistance: Month 36: number analyzed (Participants) | 217 | 522 | 937
  Had required assistance: Month 36 | 22 | 35 | 79
  Had required assistance: Month 48: number analyzed (Participants) | 203 | 466 | 852
  Had required assistance: Month 48 | 12 | 45 | 75
  Had required assistance: Month 60: number analyzed (Participants) | 82 | 180 | 369
  Had required assistance: Month 60 | 8 | 10 | 26
  Had required other assistance: Month 0: number analyzed (Participants) | 71 | 202 | 335
  Had required other assistance: Month 0 | 15 | 48 | 77
  Had required other assistance: Month 12: number analyzed (Participants) | 226 | 572 | 1011
  Had required other assistance: Month 12 | 57 | 144 | 252
  Had required other assistance: Month 24: number analyzed (Participants) | 222 | 530 | 958
  Had required other assistance: Month 24 | 57 | 135 | 241
  Had required other assistance: Month 36: number analyzed (Participants) | 217 | 523 | 936
  Had required other assistance: Month 36 | 48 | 119 | 215
  Had required other assistance: Month 48: number analyzed (Participants) | 201 | 463 | 848
  Had required other assistance: Month 48 | 49 | 119 | 211
  Had required other assistance: Month 60: number analyzed (Participants) | 82 | 180 | 367
  Had required other assistance: Month 60 | 22 | 27 | 66

20. Secondary Outcome: Health Related Productivity Questionnaire (HRPQ): Number of Participants Reporting Current Employment Status (Part Time/Full Time/Not Employed) Due to Multiple Sclerosis
Description: Participants use of healthcare resources, non-medical resources, and informal care as well as their work capacity was assessed at scheduled study visits using a modified questionnaire (HRPQ) designed to evaluate the economic impact of MS. The questionnaire addresses the following content area: participant reported data regarding employment status, work productivity, impact on household chores due to MS. Current employment status of participants (i.e. Part Time/Full Time/Not Employed) was reported in this outcome measure.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 234 | 575 | 1025
Participants
  Full time: Month 0 | 127 | 297 | 528
  Part time: Month 0 | 20 | 54 | 98
  Not employed: Month 0 | 87 | 224 | 399
  Full time: Month 12: number analyzed (Participants) | 229 | 569 | 1013
  Full time: Month 12 | 121 | 291 | 511
  Part time: Month 12: number analyzed (Participants) | 229 | 569 | 1013
  Part time: Month 12 | 20 | 53 | 104
  Not employed: Month 12: number analyzed (Participants) | 229 | 569 | 1013
  Not employed: Month 12 | 88 | 225 | 398
  Full time: Month 24: number analyzed (Participants) | 223 | 549 | 980
  Full time: Month 24 | 118 | 273 | 488
  Part time: Month 24: number analyzed (Participants) | 223 | 549 | 980
  Part time: Month 24 | 21 | 66 | 117
  Not employed: Month 24: number analyzed (Participants) | 223 | 549 | 980
  Not employed: Month 24 | 84 | 210 | 375
  Full time: Month 36: number analyzed (Participants) | 216 | 530 | 943
  Full time: Month 36 | 109 | 273 | 478
  Part time: Month 36: number analyzed (Participants) | 216 | 530 | 943
  Part time: Month 36 | 23 | 57 | 108
  Not employed: Month 36: number analyzed (Participants) | 216 | 530 | 943
  Not employed: Month 36 | 84 | 200 | 357
  Full time: Month 48: number analyzed (Participants) | 204 | 469 | 860
  Full time: Month 48 | 108 | 225 | 424
  Part time: Month 48: number analyzed (Participants) | 204 | 469 | 860
  Part time: Month 48 | 21 | 57 | 103
  Not employed: Month 48: number analyzed (Participants) | 204 | 469 | 860
  Not employed: Month 48 | 75 | 187 | 333
  Full time: Month 60: number analyzed (Participants) | 82 | 183 | 374
  Full time: Month 60 | 37 | 97 | 189
  Part time: Month 60: number analyzed (Participants) | 82 | 183 | 374
  Part time: Month 60 | 10 | 18 | 43
  Not employed: Month 60: number analyzed (Participants) | 82 | 183 | 374
  Not employed: Month 60 | 35 | 68 | 142

21. Secondary Outcome: HRPQ: Total Scheduled Working Hours and Number of Hours Missed From Work Due to Multiple Sclerosis
Description: Participants use of healthcare resources, non-medical resources, and informal care as well as their work capacity was assessed at scheduled study visits using a modified questionnaire (HRPQ) designed to evaluate the economic impact of MS. The questionnaire addresses the following content area: participant reported data regarding employment status, work productivity, impact on household chores due to MS. Data for "total scheduled working hours of participants; number of hours missed from work by participants due to MS" were reported in this outcome measure.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 153 | 380 | 675
hours
  Total scheduled working hours: Month 0: number analyzed (Participants) | 153 | 374 | 660
  Total scheduled working hours: Month 0 | 34.0 (14.6) | 32.2 (16.1) | 32.9 (16.1)
  Total scheduled working hours: Month 12: number analyzed (Participants) | 152 | 380 | 675
  Total scheduled working hours: Month 12 | 33.6 (15.4) | 32.3 (16.6) | 32.5 (16.6)
  Total scheduled working hours: Month 24: number analyzed (Participants) | 149 | 367 | 647
  Total scheduled working hours: Month 24 | 33.2 (15.5) | 30.8 (16.1) | 31.6 (16.1)
  Total scheduled working hours: Month 36: number analyzed (Participants) | 137 | 343 | 615
  Total scheduled working hours: Month 36 | 33.6 (16.4) | 33.1 (15.1) | 33.3 (15.3)
  Total scheduled working hours: Month 48: number analyzed (Participants) | 137 | 302 | 559
  Total scheduled working hours: Month 48 | 34.4 (19.7) | 31.3 (16.3) | 32.9 (17.0)
  Total scheduled working hours: Month 60: number analyzed (Participants) | 52 | 124 | 249
  Total scheduled working hours: Month 60 | 27.3 (18.9) | 31.1 (15.8) | 31.1 (16.6)
  Number of hours missed from work: Month 0: number analyzed (Participants) | 8 | 21 | 39
  Number of hours missed from work: Month 0 | 9.8 (12.1) | 15.2 (15.0) | 11.7 (12.8)
  Number of hours missed from work: Month 12: number analyzed (Participants) | 14 | 23 | 47
  Number of hours missed from work: Month 12 | 6.7 (3.6) | 10.1 (12.2) | 9.0 (10.2)
  Number of hours missed from work: Month 24: number analyzed (Participants) | 9 | 22 | 41
  Number of hours missed from work: Month 24 | 6.7 (6.1) | 10.6 (11.3) | 10.4 (10.9)
  Number of hours missed from work: Month 36: number analyzed (Participants) | 6 | 21 | 35
  Number of hours missed from work: Month 36 | 9.3 (5.9) | 24.7 (65.4) | 18.7 (50.8)
  Number of hours missed from work: Month 48: number analyzed (Participants) | 11 | 21 | 42
  Number of hours missed from work: Month 48 | 21.5 (23.1) | 37.7 (107.6) | 28.0 (77.1)
  Number of hours missed from work: Month 60: number analyzed (Participants) | 2 | 5 | 12
  Number of hours missed from work: Month 60 | 14.5 (13.4) | 13.4 (13.4) | 13.9 (13.0)

22. Secondary Outcome: HRPQ: Percentage Impact on Work Output Due to Multiple Sclerosis
Description: Participants use of healthcare resources, non-medical resources, and informal care as well as their work capacity was assessed at scheduled study visits using a modified questionnaire (HRPQ) designed to evaluate the economic impact of MS. The questionnaire addresses the following content area: participant reported data regarding employment status, work productivity, impact on household chores due to MS. Percentage impact on work output due to MS were reported in this outcome measure.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percentage impact on work output
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab (Overall)
Number analyzed (Participants) | 145 | 351 | 622
percentage impact on work output
  Month 0: number analyzed (Participants) | 145 | 349 | 622
  Month 0 | 6.2 (14.4) | 10.2 (22.3) | 8.5 (19.5)
  Month 12: number analyzed (Participants) | 138 | 351 | 622
  Month 12 | 8.7 (18.0) | 9.5 (21.5) | 9.0 (20.2)
  Month 24: number analyzed (Participants) | 137 | 335 | 596
  Month 24 | 9.9 (20.4) | 9.4 (21.2) | 9.8 (21.3)
  Month 36: number analyzed (Participants) | 128 | 316 | 571
  Month 36 | 9.2 (20.0) | 9.9 (21.3) | 9.4 (19.9)
  Month 48: number analyzed (Participants) | 129 | 279 | 525
  Month 48 | 12.2 (25.4) | 9.3 (21.7) | 9.7 (22.0)
  Month 60: number analyzed (Participants) | 43 | 115 | 231
  Month 60 | 11.7 (22.3) | 8.1 (18.9) | 9.2 (19.9)

23. Secondary Outcome: HRPQ: Total Scheduled Household Chores Hours; Number of Hours Missed From Household Chores Due to Multiple Sclerosis
Description: Participants use of healthcare resources, non-medical resources, and informal care as well as their work capacity was assessed at scheduled study visits using a modified questionnaire (HRPQ) designed to evaluate the economic impact of MS. The questionnaire addresses the following content area: participant reported data regarding employment status, work productivity, impact on household chores due to MS. Data for "total scheduled household chores hours; number of hours missed from planned household chores by participants due to MS" were reported in this outcome measure.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: Analysis was performed on efficacy population.Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants with available data for each specified category. As pre-specified, data collection and analysis for this outcome measure was done on the overall population along with 2 subgroups (DAT and IAT).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 228 | 562 | 1004
hours
  Total scheduled household chores hours: Month 0: number analyzed (Participants) | 228 | 558 | 993
  Total scheduled household chores hours: Month 0 | 9.8 (8.3) | 11.0 (11.0) | 10.8 (10.6)
  Total scheduled household chores hours: Month 12: number analyzed (Participants) | 226 | 562 | 1004
  Total scheduled household chores hours: Month 12 | 10.3 (10.1) | 11.1 (11.7) | 10.9 (11.5)
  Total scheduled household chores hours: Month 24: number analyzed (Participants) | 219 | 538 | 954
  Total scheduled household chores hours: Month 24 | 10.2 (11.6) | 10.9 (11.4) | 10.6 (11.4)
  Total scheduled household chores hours: Month 36: number analyzed (Participants) | 203 | 505 | 899
  Total scheduled household chores hours: Month 36 | 9.7 (10.2) | 11.7 (13.1) | 11.0 (12.1)
  Total scheduled household chores hours: Month 48: number analyzed (Participants) | 193 | 452 | 825
  Total scheduled household chores hours: Month 48 | 9.9 (8.9) | 10.5 (10.6) | 10.3 (10.3)
  Total scheduled household chores hours: Month 60: number analyzed (Participants) | 77 | 178 | 363
  Total scheduled household chores hours: Month 60 | 10.4 (8.7) | 11.2 (11.1) | 11.5 (12.6)
  Number of hours missed from household chores: Month 0: number analyzed (Participants) | 39 | 104 | 188
  Number of hours missed from household chores: Month 0 | 4.7 (3.3) | 6.5 (6.9) | 6.0 (5.9)
  Number of hours missed from household chores: Month 12: number analyzed (Participants) | 47 | 90 | 173
  Number of hours missed from household chores: Month 12 | 4.9 (3.5) | 6.8 (7.7) | 6.2 (6.6)
  Number of hours missed from household chores: Month 24: number analyzed (Participants) | 35 | 104 | 181
  Number of hours missed from household chores: Month 24 | 7.8 (9.0) | 7.1 (10.6) | 6.6 (9.3)
  Number of hours missed from household chores: Month 36: number analyzed (Participants) | 33 | 91 | 161
  Number of hours missed from household chores: Month 36 | 6.1 (7.4) | 7.7 (14.2) | 7.0 (11.7)
  Number of hours missed from household chores: Month 48: number analyzed (Participants) | 37 | 74 | 143
  Number of hours missed from household chores: Month 48 | 4.8 (4.3) | 6.2 (10.6) | 5.7 (8.4)
  Number of hours missed from household chores: Month 60: number analyzed (Participants) | 15 | 24 | 51
  Number of hours missed from household chores: Month 60 | 5.3 (5.2) | 5.8 (5.1) | 5.9 (5.1)

24. Secondary Outcome: HRPQ: Percentage Impact on Work Output for Household Chores Due to Multiple Sclerosis
Description: Participants use of healthcare resources, non-medical resources, and informal care as well as their work capacity was assessed at scheduled study visits using a modified questionnaire (HRPQ) designed to evaluate the economic impact of MS. The questionnaire addresses the following content area: participant reported data regarding employment status, work productivity, impact on household chores due to MS. Percentage impact on work output for household chores due to MS were reported in this outcome measure.
Time Frame: Baseline (Month 0 of LPS13649), Month 12, Month 24, Month 36, Month 48 and Month 60
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percentage impact on work output
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 212 | 531 | 947
percentage impact on work output
  Month 0 | 16.0 (23.8) | 16.4 (26.0) | 16.8 (25.8)
  Month 12: number analyzed (Participants) | 208 | 524 | 931
  Month 12 | 18.3 (27.3) | 16.6 (26.6) | 17.7 (27.5)
  Month 24: number analyzed (Participants) | 197 | 501 | 886
  Month 24 | 20.3 (28.5) | 18.5 (27.4) | 19.4 (28.1)
  Month 36: number analyzed (Participants) | 183 | 453 | 813
  Month 36 | 17.5 (25.9) | 16.5 (26.2) | 17.6 (26.6)
  Month 48: number analyzed (Participants) | 180 | 415 | 769
  Month 48 | 19.8 (28.8) | 17.0 (26.8) | 18.6 (27.7)
  Month 60: number analyzed (Participants) | 75 | 170 | 344
  Month 60 | 18.8 (28.3) | 13.1 (22.9) | 14.8 (25.0)

25. Secondary Outcome: HRPQ: Duration of Disease (in Months) Since Development of Multiple Sclerosis
Description: Participants use of healthcare resources, non-medical resources, and informal care as well as their work capacity was assessed at scheduled study visits using a modified questionnaire (HRPQ) designed to evaluate the economic impact of MS. The questionnaire addresses the following content area: participant reported data regarding employment status, work productivity, impact on household chores due to MS. Mean and standard deviation data for duration of MS disease (in months) since the start of MS development in participants was reported in this outcome measure.
Time Frame: Baseline up to end of the study (up to a maximum duration of 5.6 years)
Population: Analysis was performed on efficacy population. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. As pre-specified, data collection and analysis for this outcome measure was done on the overall population along with 2 subgroups (DAT and IAT).
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 228 | 559 | 997
months | 10.3 (4.0) | 10.2 (5.0) | 10.5 (4.5)

26. Secondary Outcome: HRPQ: Number of Participants Who Reported Impact on Work Due to Multiple Sclerosis
Description: Participants use of healthcare resources, non-medical resources, and informal care as well as their work capacity was assessed at scheduled study visits using a modified questionnaire (HRPQ) designed to evaluate the economic impact of MS. The questionnaire addresses the following content area: participant reported data regarding employment status, work productivity, impact on household chores due to MS. Number of participants who reported "Yes" as an answer to questions related to impact on work: "forced me to work part-time when I wanted to work full-time; kept me from having a job when I wanted to work full-time; kept me from having a job when I wanted to work part-time; none of the above" questions were reported in this outcome measure.
Time Frame: Baseline up to end of the study (up to a maximum duration of 5.6 years)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
Number analyzed (Participants) | 164 | 399 | 709
Participants
  My MS or treatments forced me to work part-time when I wanted to work full-time: number analyzed (Participants) | 22 | 81 | 125
  My MS or treatments forced me to work part-time when I wanted to work full-time | 22 | 81 | 125
  My MS or treatments kept me from having a job when I wanted to work full-time: number analyzed (Participants) | 32 | 88 | 168
  My MS or treatments kept me from having a job when I wanted to work full-time | 32 | 88 | 168
  My MS or treatments kept me from having a job when I wanted to work part-time: number analyzed (Participants) | 20 | 42 | 81
  My MS or treatments kept me from having a job when I wanted to work part-time | 20 | 42 | 81
  None of the above | 164 | 399 | 709

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected from the Baseline until the end of the study (up to a maximum duration of 5.6 years).
Description: Reported adverse events and death were TEAEs that is AEs that developed/worsened during the 'treatment period' (time from Baseline until the end of the study). Analysis was performed on safety population. As pre-specified, safety analysis was done on the overall population along with 2 subgroups (DAT and IAT).
Arm/Group | Delayed Alemtuzumab Treatment (DAT) | Initial Alemtuzumab Treatment (IAT) | Alemtuzumab
All-Cause Mortality (participants affected / at risk) | 0/241 | 10/598 | 11/1062
Serious Adverse Events (participants affected / at risk) | 55/241 | 133/598 | 237/1062
Other Adverse Events (participants affected / at risk) | 150/241 | 338/598 | 601/1062
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Alemtuzumab Treatment (DAT) (N=241) | Initial Alemtuzumab Treatment (IAT) (N=598) | Alemtuzumab (N=1062)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 2 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (3)
Acute Left Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 2 (2) | 4 (4)
Atrioventricular Block (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Bundle Branch Block Left (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Ventricular Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Congenital Cystic Kidney Disease (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Congenital Nail Disorder (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Foetal Chromosome Abnormality (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1)
Haematotympanum (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Autoimmune Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Autoimmune Thyroid Disorder (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Autoimmune Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Basedow's Disease (Endocrine disorders) | 2 (2) | 4 (4) | 7 (7)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Thyroid Dermatopathy (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2) | 1 (2)
Endocrine Ophthalmopathy (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Exophthalmos (Eye disorders) | 1 (2) | 0 (0) | 1 (2)
Eyelid Ptosis (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Optic Ischaemic Neuropathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital Oedema (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Intestinal Ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Obstructive Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Pancreatitis Chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (3)
Catheter Site Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Complication Associated With Device (General disorders) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2) | 2 (2)
Drug Intolerance (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Sudden Death (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 4 (4)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Immune Reconstitution Inflammatory Syndrome (Immune system disorders) | 1 (2) | 0 (0) | 1 (2)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Abscess Rupture (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 3 (7) | 4 (8)
Cellulitis Staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Clostridium Difficile Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal Bacterial Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Herpes Zoster Infection Neurological (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infected Bite (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infected Lymphocele (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Klebsiella Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Localised Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neonatal Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Osteomyelitis Acute (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4) | 9 (10)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Pneumonia Streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Scrotal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (3) | 5 (7)
Septic Shock (Infections and infestations) | 0 (0) | 3 (3) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 2 (3) | 4 (4) | 9 (10)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Uterine Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 3 (3)
Brain Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Burns Third Degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Face Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 2 (3)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Induced Abortion Failed (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 1 (3)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skull Fractured Base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Ulna Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Antiphospholipid Antibodies Positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
Human Papilloma Virus Test Positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic Ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 3 (4)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Joint Contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 2 (4)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brenner Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Cutaneous T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Gallbladder Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3)
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Laryngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Lung Squamous Cell Carcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Malignant Neoplasm Of Unknown Primary Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Ovarian Germ Cell Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 5 (5)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Limbic Encephalitis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Lumbosacral Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Multiple Sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple Sclerosis Relapse (Nervous system disorders) | 6 (6) | 18 (30) | 30 (43)
Optic Neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Partial Seizures (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Post Herpetic Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Postural Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Resting Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Uhthoff's Phenomenon (Nervous system disorders) | 3 (3) | 5 (5) | 9 (9)
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (5) | 6 (7) | 11 (15)
Anembryonic Gestation (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 0 (0) | 1 (2)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1)
Foetal Distress Syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Hellp Syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Missed Labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1)
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (3) | 4 (4) | 7 (8)
Prolonged Labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Behaviour Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Completed Suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 4 (4)
Depression Suicidal (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Drug Abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Substance-Induced Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 2 (2) | 2 (3) | 4 (5)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Lupus Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (3) | 2 (2) | 5 (7)
Renal Colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal Injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (2)
Cervical Dysplasia (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 5 (5)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 2 (3)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral Artery Thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Alemtuzumab Treatment (DAT) (N=241) | Initial Alemtuzumab Treatment (IAT) (N=598) | Alemtuzumab (N=1062)
Nausea (Gastrointestinal disorders) | 13 (13) | 18 (18) | 37 (37)
Fatigue (General disorders) | 15 (17) | 19 (19) | 43 (45)
Bronchitis (Infections and infestations) | 14 (17) | 44 (54) | 67 (81)
Herpes Zoster (Infections and infestations) | 15 (16) | 29 (35) | 50 (57)
Influenza (Infections and infestations) | 13 (13) | 25 (28) | 48 (55)
Nasopharyngitis (Infections and infestations) | 34 (60) | 73 (112) | 129 (204)
Sinusitis (Infections and infestations) | 11 (11) | 34 (45) | 57 (71)
Upper Respiratory Tract Infection (Infections and infestations) | 27 (29) | 50 (73) | 96 (123)
Urinary Tract Infection (Infections and infestations) | 37 (56) | 78 (143) | 151 (271)
Fall (Injury, poisoning and procedural complications) | 15 (20) | 27 (34) | 54 (74)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (27) | 39 (45) | 69 (86)
Back Pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 30 (34) | 62 (68)
Headache (Nervous system disorders) | 37 (52) | 67 (87) | 125 (164)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 14 (23) | 39 (46) | 63 (86)
Depression (Psychiatric disorders) | 13 (13) | 25 (26) | 43 (45)
Insomnia (Psychiatric disorders) | 16 (17) | 29 (32) | 57 (62)
Rash (Skin and subcutaneous tissue disorders) | 13 (16) | 26 (34) | 51 (64)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT02255656/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT02255656/SAP_001.pdf